CLINICAL TRIAL: NCT05509920
Title: Assessment of Arresting Root Surface Caries After the Application of PRG Bioactive Varnish Versus SDF Varnish Over a Period of 1 Year Follow up
Brief Title: Assessment of Arresting Root Surface Caries After the Application of PRG Bioactive Varnish
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Sayed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Giomer based barrier coat
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Root Caries
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with root carious lesions will be treated by SDF varnish (Active Comparator): Silver diamine fluoride (SDF) contains high concentrations of silver and fluoride ions, which prevents and arrests root caries, as well as dentin caries in the primary teeth of young children. Unlike other fluoride products that mainly reduce the formation of new carious lesions, 38% SDF is an effective agent that can efficiently arrest the carious process, remineralize the decayed dental tissues, and protect the tooth structure against the for-mation of new caries lesions. The use of SDF can result in more caries-resistant tooth structures.
  Interventions: Other: S-PRG barrier coat
- patients with root carious lesions will be treated by PRG barrier coat. (Experimental): PRG barrier coat is a Giomer varnish from Shofu. It is a light cured Surface-partially reacted glass (S-PRG) filler particles with a multifunctional glass core embedded in a resin matrix. It has an immediate and long lasting effect. The (S-PRG) favors the re-lease of fluoride ions and its recharging that aid in remineraliza-tion and protection of the tooth structure in a way similar to the glass ionomer. The fluoride ions aid in the neutralization of the acidity of the oral cavity and decrease the plaque accumulation
  Interventions: Other: S-PRG barrier coat

INTERVENTIONS:
Other: S-PRG barrier coat — S-PRG filler was the best composition of compressive strength and F- and B release acid buffering capacity. It was found to be the most promising for use as a novel cement.

SUMMARY:
Guidelines proved that arresting and remineralization of the root surface caries is better than weakening the tooth structure and restoring it. Manufacturer claims that PRG Barrier Coat effectively treats dental hypersensitivity by providing immediate and long-lasting relief. Also has the effect of eliminating the activity and sur-vival of pathogenic bacteria and hardening the dentin tissue of the affected areas.

DETAILED DESCRIPTION:
A light-cured varnish with extended protection time of up to 6 months, PRG barrier coat incorporates proprietary GIOMER tech-nology, "Surface Pre-Reacted Glass" for high fluoride release and re-charge, continuous release of fluoride, strontium, boron, sodium, aluminum, and zinc, acid neutralization and anti-plaque benefits with excellent self-adhesive abilities. The new material could be an alter-native to SDF varnish in root caries arrest to overcome its unfavor-able color and taste.

Products containing S-PRG fillers have been developed in a wide variety of areas such as tooth surface coating materials, seal-ants, restoration resins and dentifrices. The use of these materials is also expected to have the effect of improving the properties of enamel. In this seminar, we will introduce a new caries prevention using S-PRG filler The eluted ions from the S-PRG filler containing materials exhibit various functions, such as prohibition of biofilm attachment, anti-demineralization, remineralization, modification of apatite crystal, and acid-buffering effect. Each ion was confirmed its function. Par-ticularly, Strontium, Borate and Fluoride ions were involved during calcium phosphate nucleation to form modified nano-hydroxyapatite. The acid buffering effect was shown with the borate ion. As the results of those effects of ions, the various materials with S-PRG technology were proven to con-tribute to increase the acid resistance and the caries prevention.

ELIGIBILITY:
Inclusion Criteria:

* Teeth with primary root surface caries (active dentin carious le-sions)
* Teeth with gum recession.
* Teeth are vital according to pulp-sensitivity tests.
* Controlled gingival or periodontal conditions.

Exclusion Criteria:

* Retained deciduous teeth; as the research is targeting only per-manent teeth.
* Teeth with previous restorations which may add another varia-ble to the study (type of old restorative material, extent of re-current caries).
* Spontaneous pain or prolonged pain after sensitivity tests (cold and electrical tests) indicating irreversible pulpitis.
* Negative sensitivity tests, periapical radiolucencies, and sensi-tivity to axial or lateral percussion indicating pulp necrosis.
* Teeth presenting external or internal resorption, with adverse pulpal reactions which may affect the outcome of the study.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of caries arrest | one year
  Evaluation of caries arrest by visual tactile evaluation. (mean number of arrested carious lesions that become hard, smooth and free from plaque post application of both SDF and S-PRG varnishes).

IPD SHARING:
Plan to Share IPD: Undecided